CLINICAL TRIAL: NCT03641846
Title: "Low-intensity Shockwave Therapy (LiST) for the Treatment of Mild and Mild-to-moderate Vasculogenic Erectile Dysfunction: a Randomized Placebo Controlled Two-parallel Arms Trial, Comparing 6 Sessions, With Daily Tadalafil 5mg vs Placebo"
Brief Title: Low-intensity Shockwave Therapy (LiST) for the Treatment of Mild and Mild-to-moderate Vasculogenic Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, Chairman, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10672/2018
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Erectile Dysfunction; Low Intensity Shockwave Therapy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LiST + 5mg Tadalafil Group (Active Comparator): All patients will receive shockwave treatment (6 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), twice per week (total of 3 weeks) without treatment interval. Starting at first LiST session and finishing one week after final LiST session, subjects will receive for 4 weeks daily Tadalafil 5mg. Total treatment period = 4 weeks.
  Interventions: Other: DornierAries2 LiST device + 5 mg Tadalafil
- LiST+Placebo Group (Placebo Comparator): All patients will receive shockwave treatment (6 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), twice per week (total of 3 weeks) without treatment interval. Starting at first LiST session and finishing one week after final LiST session, subjects will receive for 4 weeks daily placebo pill. Total treatment period = 4 weeks.
  Interventions: Other: DornierAries2 LiST device + Placebo Pill

INTERVENTIONS:
Other: DornierAries2 LiST device + 5 mg Tadalafil — All patients will receive shockwave treatment (6 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), twice per week (total of 3 weeks) without treatment interval. Starting at first LiST session and finishing one week after final LiST session, subjects will receive for 4 weeks daily Tadalafil 5mg. Total treatment period = 4 weeks
  Arms: LiST + 5mg Tadalafil Group
Other: DornierAries2 LiST device + Placebo Pill — All patients will receive shockwave treatment (6 sessions for all subjects, 5000 shockwaves at each session, at energy level 7), twice per week (total of 3 weeks) without treatment interval. Starting at first LiST session and finishing one week after final LiST session, subjects will receive for 4 weeks daily Placebo pills. Total treatment period = 4 weeks.
  Arms: LiST+Placebo Group

SUMMARY:
This is a randomized, double-blind, 2 parallel arms clinical trial. All patients will be PDE5I users/responders. After 1 month wash-out period, ED patients will be screened, in order to randomize 50 men with vasculogenic ED with primary objective to examine the efficacy of LiST using Aries2 device.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 40-70 years.
3. Sexually active in a stable, heterosexual relationship of more than three months duration.
4. Presence of Erectile Dysfunction for at least 6 months.
5. At Screening, diagnosed as Vasculogenic erectile dysfunction based on sexual history
6. PDE5i users and report some or good response to PDE5i. Last reported PDE5i use must be within 30 days of Screening Visit.
7. Agree to suspend all other ED therapies, except the assigned study treatments, for the duration of the study.
8. Agree to attempt sexual intercourse at least 4 times during the last 4 weeks prior to Visit 2/Randomization, 1-month Follow Up, 3-month Follow-Up and 6-month Follow-Up without being under the influence of alcohol or recreational drugs. Agree to document the outcome using the Sexual Encounter Profile (SEP) diary.
9. IIEF-EF score 17-25 at Visit 2 (after PDE5i washout)
10. At Visit 2 (after PDE5i washout), SEP Q2, "Were you able to insert your penis into your partner's vagina?" answered "YES" 50% - 100% of the time.
11. At Visit 2, SEP Q3, "Did your erection last long enough for you to have successful intercourse?" answered "YES" < 100% of the time.

Exclusion Criteria:

1. Previous major pelvic surgery or pelvic trauma that could impact erectile function, such as radical prostatectomy, radical cystectomy, rectal surgery. Patients with previous TURP surgery without sequelae of iatrogenic ED, may be included.
2. Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, grafting.
3. Previous history of priapism or penile fracture
4. Previous radiation therapy to pelvis.
5. Abnormal serum testosterone level defined as a value lower than 300 ng/dL (indicative of untreated hypogonadism), or greater than 1197 ng/dL.
6. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
7. ED due primarily to psychogenic factors.
8. Peyronie's Disease or penile curvature that negatively influences sexual activity.
9. Patients with cardiac or non-cardiac electrical devices implanted.
10. Open wounds, or any anatomical or neurological abnormalities in the treatment area.
11. Uncontrolled diabetes mellitus with glucose >200 mg/dL (once or more times/week during the last month prior to recruitment, or during screening blood test).
12. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's Disease.
13. Refusal to suspend alternative ED therapy for duration of study. Subjects who are using Tadalafil as a treatment for BPH (Benign Prostatic Hyperplasia) will also be excluded.
14. Men deemed not healthy enough to participate in sexual activity.
15. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
16. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
17. Known allergy to ultrasound gel.
18. History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
19. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using SSRI or psychotropic medications e.g., Citalopram (Celexa), Escitalopram (Lexapro, Cipralex), Paroxetine (Paxil, Seroxat), Fluoxetine (Prozac), Fluvoxamine (Luvox, Faverin),Sertraline (Zoloft, Lustral), Clonazepam (Klonopin), Alprazolam (Xanax), Aripiprazole (Ambilify), Clozapine (Clozaril), Risperidone (Risperdal), Quetiapine (Seroquel), Olanzapine (Zyprexa) are also excluded.
20. Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.
21. History of adverse events in response to tadalafil, which would prevent the patient from being blinded to his group allocation, and/or prevent patient compliance to the study protocol.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Change in the Erectile Function domain score of the International Index of Erectile Function (IIEF-EF) | baseline and 12-week follow-up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)

SECONDARY OUTCOMES:
Change in the Erectile Function domain score of the International Index of Erectile Function (IIEF-EF) | baseline and 4-week follow-up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
Change in the Erectile Function domain score of the International Index of Erectile Function (IIEF-EF) | baseline and 24-week follow-up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 4-week follow-up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 12-week follow-up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Change in Sexual Encounter Profile Question 3 (SEP3) score | baseline and 24-week follow-up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported.The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4). SEP 3 exact question is "Did your erection last long enough for you to have successful intercourse?"
Number of patients with treatment related adverse events | 28 weeks
  Potential treatment related adverse events after the first LI-ESWT session and during the 6 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases, Thessaloniki, Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided